CLINICAL TRIAL: NCT05667142
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 3 Study to Evaluate the Safety, Tolerability, and Efficacy of XEN1101 as Adjunctive Therapy in Primary Generalized Tonic-Clonic Seizures
Brief Title: A Study to Evaluate XEN1101 as Adjunctive Therapy in Primary Generalized Tonic-Clonic Seizures
Acronym: X-ACKT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPF-010-303; 2022-502286-16-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Primary Generalized Tonic-Clonic Seizures
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- XEN1101 25 mg/day (Experimental): XEN1101 25 mg/day
  Interventions: Drug: XEN1101
- XEN1101 15 mg/day (Experimental): XEN1101 15 mg/day
  Interventions: Drug: XEN1101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN1101 — XEN1101 capsules
  Other Names: Azetukalner
  Arms: XEN1101 15 mg/day; XEN1101 25 mg/day
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the clinical efficacy, safety, and tolerability of XEN1101 administered as adjunctive treatment in primary generalized tonic-clonic seizures (PGTCS).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the clinical efficacy, safety, and tolerability of XEN1101 administered as adjunctive treatment in subjects diagnosed with generalized epilepsy and experiencing probable or possible PGTCS (with or without other subtypes of generalized seizures), and taking 1 to 3 anti-seizure medications (ASMs). Eligible subjects will be randomly assigned 1:1 to XEN1101 or placebo: subjects aged ≥ 18 years will receive XEN1101 25 mg or placebo, and subjects aged ≥12 years and <18 years will receive either XEN1101 15 mg, 25 mg, or placebo. Randomization will be stratified based on region, age group, and background use of CYP3A4-inducer ASMs. Eligible subjects will have up to 9.5 weeks durations to assess the baseline frequency of seizures, followed by a double-blind treatment period (DBP) where subjects will receive 12 weeks of blinded treatment. During the DBP, subjects will be instructed to orally take XEN1101 or placebo once daily with an evening meal.

Subjects who complete the 12-week DBP will have the opportunity to enroll in a separate open-label-extension (OLE) study for continued treatment with XEN1101. Subjects who do not enroll in the OLE will enter an 8 week post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is properly informed of the nature and risks of the study and gives informed consent in writing prior to entering the study (for adult subjects) and for adolescent subjects parent/legal guardian and subject gives informed consent or assent in writing prior to entering the study.
2. Subject is ≥12 years of age with a BMI ≤40 kg/m2 at Visit 1.
3. Subject must have had adequate trials of at least 2 ASMs, which were given (and tolerated) at adequate therapeutic doses, without achieving sustained seizure freedom.
4. Subject has probable or possible PGTCS (with or without other subtypes of generalized seizures) for ≥1 year, in the setting of generalized epilepsy according to the International League Against Epilepsy 2017 classification criteria, and subject is approved by The Epilepsy Study Consortium (TESC).
5. Subject is on a stable dose of 1 to 3 allowable current ASMs for at least 1 month prior to screening (Visit 1), during screening/baseline, and throughout the DBP.
6. Subject is able to keep accurate seizure diaries.

Exclusion Criteria:

1. Subject has had status epilepticus within the 12 months prior to Visit 1.
2. Subject has history of repetitive seizures within the 12-month period preceding Visit 1 where the individual seizures cannot be counted.
3. Subject has a history of non-epileptic psychogenic seizures.
4. Subject has a concomitant diagnosis of focal-onset seizures (FOS).
5. Subject has presence or history of a developmental and epileptic encephalopathy, including Lennox-Gastaut syndrome.
6. Subject has seizures secondary to drug or alcohol use, ongoing infection, neoplasia, demyelinating disease, degenerative neurological disease, metabolic illness, progressive structural lesion, encephalopathy, or progressive central nervous system (CNS) disease.
7. Subject has history of neurosurgery for seizures <1 year prior to Visit 1, or radiosurgery <2 years prior to Visit 1.
8. Subject has schizophrenia and other psychotic disorders (eg, schizophreniform disorder, schizoaffective disorder, psychosis not otherwise specified), bipolar disorder, obsessive-compulsive disorder, or another serious mental health disorder. Subject has uncontrolled unipolar major depression where changes in pharmacotherapy are needed or anticipated during the study.
9. Subject has any clinically significant laboratory abnormalities or clinically significant abnormalities on prestudy physical examination, vital signs, or ECG that, in the judgment of the investigator, indicate a medical problem that would preclude study participation, including but not limited to:

   a. History or presence of long QT syndrome; QTcF >450 msec at baseline; family history of sudden death of unknown cause.
10. Any personal circumstance that, in the opinion of the investigator, prevents adherence to the protocol.

The criteria to be eligible for randomization are:

1. During the last 56 days of the baseline period that preceded the randomization visit (Visit 2), subject must have had a sufficient documented seizure frequency of PGTCS, including ≥1 PGTCS during each of the first and second 4-week periods preceding randomization.
2. Seizure diary was completed a minimum of 80% of all days (ie, ≥45 days) during the last 56 days of the baseline period that preceded randomization as evidence of adequate compliance.
3. Subject did not change dose of, stop, or initiate any new ASM(s) during the baseline period and plans on maintaining a stable dose of ASM(s) during the DBP.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Median percent change (MPC) in monthly (28 days) PGTCS frequency | Baseline through DBP (Week 12)
  Median percent change (MPC) in monthly (28 days) PGTCS frequency from baseline through the DBP for XEN1101 versus placebo.

SECONDARY OUTCOMES:
Proportion of subjects | Baseline through DBP (Week 12)
  Proportion of subjects experiencing ≥50% reduction in monthly (28 days) PGTCS frequency from baseline through the DBP for XEN1101 versus placebo.
Proportion of subjects | Baseline through Week 12
  Proportion of subjects experiencing PGTCS freedom from baseline through the DBP for XEN1101 versus placebo.

OTHER OUTCOMES:
Incidence of adverse events | From Screening Through to 56 Days Post-Final Dose
  To assess the safety and tolerability of XEN1101 in subjects with PGTCS (e.g., adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (137):
- United States (58):
  - University of Alabama - Strada Patient Care Center, Neurology, Mobile, Alabama
  - Xenoscience, Phoenix, Arizona
  - University of Arizona - Health Science Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Brain Science Research Institute, Los Angeles, California
  - University of California, Irvine - Health Neurology Services, Orange, California
  - University California, Davis Clinical & Translation Science Center Clinical Research (CCRC), Sacramento, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Serenity Research Center, LLC, Miami, Florida
  - Research Institute of Orlando, LLC, Orlando, Florida
  - Panhandle Research and Medical Clinic, Pensacola, Florida
  - Medsol Clinical Research Center Harbor Professional Centre, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Encore Medical Research of Weston, LLC, Weston, Florida
  - Emory Brain Health Center, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Georgia Neurology & Sleep Medicine Associates, Suwanee, Georgia
  - Hawaii Pacific Neuroscience, Comprehensive Epilepsy Center, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - University of Kentucky Albert B. Chandler Hospital (UK Healthcare), Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Medstar Georgetown University Hospital, Clinton, Maryland
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Michigan State University Department of Neurology, East Lansing, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Saint Louis University Medical School, St Louis, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Dent Neurosciences Research Facility, Amherst, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Five Towns Neurology, Woodmere, New York
  - Atrium Health, Charlotte, North Carolina
  - Onsite Clinical Solutions, LLC, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Summa Health Clinical Research Center, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Comprehensive Epilepsy Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - ANESC Research, El Paso, Texas
  - UTHealth Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - University of Washington, Regional Epilepsy Center at Harborview Medical Center, Seattle, Washington
  - Advocate Aurora Research institute, St. Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (4):
  - Hospital General de Agudos J.M. Ramos Mejia, Buenos Aires
  - STAT Research S.A., Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Sanatorio del Sur S.A, San Miguel de Tucumán
- Australia (6):
  - Southern Neurology, Kogarah, New South Wales
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - The Alfred Hospital, Melbourne, VC
  - Austin Health Pharmacy Clinical Trials, Heidelberg, Victoria
  - St Vincent's Hospital Melbourne, Clinical Neurosciences, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville
- Austria (4):
  - University Hospital Innsbruck, Innsbruck
  - Universitaetsklinik fuer Kinder, Linz
  - Universitätsklinik für Neurologie, Salzburg
  - Universitätsklinik für Neurologie, Medizinische Universität Wien, Vienna
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Bulgaria (3):
  - Multiprofile hospital for active treatment Puls AD, Blagoevgrad
  - MHATNP 'Sveti Naum' EAD, Sofia
  - First University Multiprofile Hospital for Active Treatment Sofia Sv. Joan Krastitel, Sofia
- Canada (4):
  - Center for Neurologic Research, Lethbridge, Alberta
  - Children and Women's Health Centre of BC (BC Children's Hospital), Vancouver, British Columbia
  - London Health Sciences Center, London, Ontario
  - Le Centre Hospitalier de l'Universite' de Montreal (CHUM), Montreal, Quebec
- Centro de investigación Clinica UC-CICUC, Santiago, Chile
- Croatia (3):
  - Clinical Hospital Center Osijek, Osijek
  - Clinical Hospital Center Rijeka, Rijeka
  - University Hospital Center Zagreb, Zagreb
- Fakultni nemocnice v Motole Neurologicka klinika 2. LF UK a FN Motol, Prague, Czechia
- France (5):
  - CHU de Lille, Hôpital Roger Salengro - Neurophysiologie clinique, Lille
  - Hopital Neurologique Pierre Wertheimer, Hospices Civils de Lyon, Lyon
  - Hôpital Fondation A. de Rothschild, Paris
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (10):
  - Universitätsklinikum Aachen, Aachen
  - Vivantes Humboldt Klinikum, Berlin
  - Bethel Epilepsy Centre, Bielefeld
  - Universitätsklinikum Frankfurt, Frankfurt
  - Epilepsiezentrum im Neuozentrum, Freiburg im Breisgau
  - Philipps-Universität Marburg, Marburg
  - Klinikum der Universität München, München
  - Epilepsiezentrum Kleinwachau gemeinnützige GmbH, Radeberg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Israel (4):
  - Hadassah University Medical Center, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Ancona, Ancona
  - Università Degli Studi Gabriele d'Annunzio Di Chieti, Chieti
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedalo Pediatrico Bambino Gesu, Roma
  - Policlinico Umberto I, Roma
- Mexico (3):
  - Grupo Medico Camino SC, Mexico City
  - Human Science Research Trials S. de R.L. de C.V., Mexico City
  - Neurociencias Estudios Clínicos S.C, Sinaloa
- Kempenhaeghe, Heeze, Netherlands
- Poland (5):
  - Centrum Medyczne Neuromed, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o.o., Gdansk
  - Novo-Med Zielinski I Wspolnicy Sp. J., Katowice
  - NZOZ Neuromed M. i M., Lublin
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól
- Portugal (7):
  - Centro Hospitalar Universitário de Coimbra (CHUC), Coimbra
  - Hospital da Senhora da Oliveira, Guimarães
  - Centro Hospitalar Lisboa Ocidental, Hospital Egas Moniz, Lisbon
  - Centre Hospitalar Universitario de Lisboa Norte (CHULN), Lisbon
  - Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - Centro Hospitalar Universitário de Santo António, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, Santa Maria da Feira
- Spain (5):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Vithas Madrid La Milagrosa, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Clinico Viña del Mar, Valparaíso
- United Kingdom (6):
  - University Hospital of Wales, Cardiff, Wales
  - Mid Yorkshire Hospitals NHS Trust, Wakefield, West Yorkshire
  - St George's University Hospitals NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - John Radcliffe Hospital, Oxford
  - Salford Royal NHS Foundation Trust - Greater Manchester Neuroscience Centre (GMNC), Salford

IPD SHARING:
Plan to Share IPD: No